CLINICAL TRIAL: NCT04857203
Title: The Role of Vitamin D in Predicting Response to Neoadjuvant Therapy in Patients With Rectal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Cihad Tatar, Associate Professor, Istanbul Training and Research Hospital
Other Study IDs: 2767
Record Dates: First submitted 2021-04-21; First posted 2021-04-23 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Rectal Cancer; Stage III Rectal Cancer
Keywords: rectal cancer; neoadjuvant; vitamin D
MeSH Terms: conditions — Rectal Neoplasms | interventions — Vitamin D Response Element

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Low levels of Vitamin D
  Interventions: Diagnostic Test: Vitamin D
- Group 2: High levels of Vitamin D
  Interventions: Diagnostic Test: Vitamin D

INTERVENTIONS:
Diagnostic Test: Vitamin D — Vitamin D levels will be measured for the patients undergoing neoadjuvant therapy in patients with locally advanced rectal cancer

SUMMARY:
It has been reported that better local control is achieved and sphincters are preserved at a higher rate with curative resections performed after neoadjuvant chemoradiotherapy in patients with locally advanced rectal cancers. In addition, it has been reported that local recurrence is reduced and survival is prolonged in patients with complete pathological response to neoadjuvant therapy. Therefore, the importance of predicting patients with pathological complete response has increased.

It has been reported that data obtained from PET-CT scans and clinical information such as tumor size, T stage, and N stage may be useful in predicting the response to neoadjuvant therapy in patients with locally advanced rectal cancer.

Consideration of blood biomarkers in predicting neoadjuvant response can be a very attractive option. Because samples are easily collected, relatively inexpensive to measure, and contain information about different aspects of tumor biology. There are a limited number of blood biomarkers such as CEA and IL-6 that have been studied in the literature.

Experimental studies show that vitamin D suppresses inflammation and protects against cancer by triggering differentiation. In 1980, Cedric and Frank Garland stated for the first time that vitamin D may affect the survival of the patient after the diagnosis of colorectal cancer. In later studies, a positive relationship was reported between the serum level of 25-hydroxyvitamin D - 25 (OH) D and survival rates for colorectal cancer, breast and prostate cancer. In addition, 25 (OH) D serum concentration has been shown to be inversely related to colorectal cancer progression.

In the light of all these information, the role of serum vitamin D levels before neoadjuvant treatment in predicting pathological response in patients with rectal cancer is investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

* • All patients with locally advanced rectal cancer

Exclusion Criteria:

* • below 18 years old

  * patients who did not received neoadjuvant therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with locally advanced rectal cancer
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
The Role of Vitamin D in response to neoadjuvant therapy for the patients with locally advanced rectal cancer | 8 weeks
  The Role of Vitamin D in Predicting Response to Neoadjuvant Therapy in Patients with Rectal Cancer Vitamin D levels will be measured for all the patients just before the neoadjuvant therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Training and Research Hospital, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided